CLINICAL TRIAL: NCT04975126
Title: Computer-based Tutorial as Supportive Means to Enhance Quality and Efficiency of the Informed Consent Process for Cataract Surgery: an Exploratory Study
Brief Title: Computer-based Tutorial as Supportive Means to Enhance the Informed Consent Process for Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CatInfo
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Cataract
Keywords: Cataract surgery; informed consent process; patient education
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CatInfo tool + Face-to-face discussion with physician (Experimental): audio-visual presentation (CatInfo tool) before face-to-face informed-consent discussion with the physician
  Interventions: Other: CatInfo tool
- Face-to-face discussion with physician only (No Intervention): face-to-face informed-consent discussion with the physician only

INTERVENTIONS:
Other: CatInfo tool — Presentation about cataract surgery
  Arms: CatInfo tool + Face-to-face discussion with physician

SUMMARY:
To assess whether a computer-based tutorial as supportive means enhances quality and efficiency of the informed consent process for cataract surgery focussing on the patients' attitude before and after surgery.

DETAILED DESCRIPTION:
Informing the patient and obtaining informed consent is one of the major duties physicians perform before starting a medical treatment. The requirements concerning the informed consent process are high. The amount of information needed to be explained to the patient is growing, as procedures get more complex and the number of treatment options increase.

The CatInfo tool is a computer-based tutorial about cataract and cataract surgery run on a handheld device with headphones and presented in an audio-visual fashion. The patient gives feedback after each chapter using a traffic light system to ensure that the content has been understood (green - content understood, ready to continue; yellow - questions that require discussion with the physician and red - repetition of the module required). A printout that summarizes what the patient has selected after each chapter immediately tells the physician which topics have been poorly understood or were unclear.

It has been shown in a randomized triple-masked study that patients using the CatInfo tool were significantly better informed than patients only having a face-to-face interview. Satisfaction with the tool was high. This present study has the goal to assess the patients' attitude before and after surgery using validated questionnaires (decisional conflict scale, decision regret scale) as well as knowledge. Patients scheduled for their first eye cataract surgery are randomly allocated to two groups, receiving standard face-to-face informed consent (control group) or additionally using the interactive CatInfo tool (study group). Scores between the groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Age 18 and older
* First eye to be operated
* No previous ophthalmic surgery
* written informed consent to participation in the study

Exclusion Criteria:

* Visual acuity of less than 0.1 Snellen in the worse eye
* Severe hearing loss
* Inability to use touch screen device (e.g. severe tremor, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-04-09 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Decisional conflict scale score | Day of pre-assessment visit (1 week before surgery)
  To assess the decisional confidence after the face-to-face informed consent discussion patients are asked to complete the decisional conflict scale questionnaire. In this study it is calculated as decisional confidence, where 0 represents the lowest decisional confidence and 100 the highest.
Decision regret scale score | 1 month after surgery
  One month after surgery the patients' satisfaction with their decision is evaluated with the decision regret scale (DRS) questionnaire via telephone interview. A score of 0 means no regret, a score of 100 high regret.
Number of correctly answered questions assessing knowledge | Day of pre-assessment visit (1 week before surgery)
  To assess the knowledge concerning cataract surgery patients are asked to complete a multiple-choice questionnaire concerning cataract surgery. The number of correctly answered questions are summed up. The scale ranges from a minimum of 0 points to a maximum of 19 points. The more points the better the patient's knowledge about cataract and cataract surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, MBA, Principal Investigator — Vienna Institute for Research in Ocular surgery (VIROS), Vienna, Austria
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

REFERENCES:
- [Derived] Ullrich M, Findl O, Kefer K, Doller B, Varsits R, Hienert J, Hirnschall N. An evaluation of the efficacy of a supplemental computer-based tutorial to enhance the informed consent process for cataract surgery: an exploratory randomized clinical study. BMC Ophthalmol. 2022 Nov 11;22(1):430. doi: 10.1186/s12886-022-02652-z. PMID 36368980